CLINICAL TRIAL: NCT04809532
Title: Analgesic Efficacy of Trans Abdominis Plane Block in Women Undergoing Cesarean Section: a Randomized Study.
Brief Title: Trans Abdominis Plane (TAP) Block in Patients With Cesarean Section
Acronym: TAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, Principal Investigator, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1506/ERC/Training
Record Dates: First submitted 2021-03-08; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Analgesia; Cesarean Section Complications
Keywords: Transverse abdominis plane block; cesarean section; postoperative use of opioids
MeSH Terms: conditions — Agnosia | interventions — Dental Occlusion; Bupivacaine; Tramadol

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Transverse abdominis plane (TAP ) block via 20ml 0.25% bupvicaine on both sides of midline will be given at end of surgery
  Interventions: Procedure: Transverse abdominis plane (TAP) block; Drug: Bupivacain; Drug: Tramadol
- Group B (No Intervention): At the end of surgery, no additional intervention will be done.

INTERVENTIONS:
Procedure: Transverse abdominis plane (TAP) block — Ultrasound guide bilateral TAP block at end of cesarean section
  Arms: Group A
Drug: Bupivacain — 20ml 0.25% bupvicaine
  Arms: Group A
Drug: Tramadol — intravenous tramadol
  Arms: Group A

SUMMARY:
Objective: To compare Trans Abdominis Plane block in providing post cesarean analgesia with control group, in terms of mean postoperative use of Opioids.

Study design: Randomized controlled trial. Place and duration Department of Anesthesiology, Combined Military Hospital, Sargodha, 25th February 2021 to 25th April 2021.

Materials and methods: A total of 60 female patients, who are planned to undergo elective c section and aged between 20-45 will be selected randomly and divided into two groups ( A and B) with 30pts each group. In Group A, at the end of surgery, TAP block will be given with 20ml of 0.25%bupvicaine via ultrasound guided sub-costal approach on both sides of midline. Time of TAP block will be recorded as time 0. Our outcomes will be: mean postoperative consumption of opioids and VAS score within 24hrs of surgery. Independent t test will be used to compare group A and B in terms of mean usage of tramadol within 24hrs of surgery. P value <0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
Analgesic efficacy of trans abdominis plane block in women undergoing Cesarean section: a randomized controlled trial.

Introduction:

Cesarean section is considered as one of the most commonly performed surgery worldwide. Based on the data from 121 countries, the trend analysis showed that between 1990 and 2014, the global average CS rate increased 12.4% (from 6.7% to 19.1%) with an average annual rate of increase of 4.4%.Its incidence in 2010 and 2013 was 41.9% and 48% respectively which was contrary to the rate of C/S recommended by the World Health Organization as fifteen percent for year 2014 .Just like all other major abdominal surgeries, c section comes with severe postoperative pain ,which if not managed properly can not only leads to prolonged immobility and its associated adverse effects but can also affect mother-baby bonding, care of baby, breast feeding and may lead to chronic pain and post-partum depression Multiple modalities are available for managing this post cesarean pain. Mostly systemic opioids are used but they are often associated with a number of undesirable side effects such as nausea, vomiting, pruritus, constipation, and respiratory depression,sedation.Other than opoids, systemic NSAIDS such as ketorolac, acetoaminophen are also used but alone they may be insufficient to treat post cesarean pain. Other analgesic options currently being used include local anesthetic techniques (local anesthetic infiltration, neuraxial blocks) acetaminophen , cyclooxygenase-2-specific inhibitors as well as analgesic adjuncts such as steroids, ketamine and α-2 agonists such as clonidine.

Neruoaxial anesthesia such as lumbar or thoracic epidurals are also used but because of constant and strict monitoring ,they are not considered economical for patients as well as for hospitals. With recent advancements in regional anesthesia, some regional blocks are now being utilized for postoperative pain relief in c sections such as TAP blocks but their use is still limited because of nonavailability of sufficient data.

Transversus abdominis plane (TAP) block provides analgesia by blocking nerves in anterior abdominal wall through introduction of a long-acting local anesthetic solution between the internal oblique and transversus abdominis muscles. Its use in c section is still limited ,but is considerd to be increased in future as is now been shown by several studies .

One of these studies is done by Uma Srivastava and collegues which showed that cumulative tramadol usage during first 24 h after surgery was significantly reduced in women given TAP block in comparison to control group C (75 ± 22 vs. 168 ± 45 mg in groups B and C, respectively, P < 0.0001.

As no local study is available and in the light of above mentioned studies, we proposed that with bilateral TAP block after c section you can provide better analgesia and improve patient's quality of life in postoperative period by reducing opoid usage and its associated side effects .

OBJECTIVE:

To compare TAP block in providing post cesarean analgesia with control group, in terms of mean reduction in postoperative use of opoids.

OPERATIONAL DEFINITIONS:

TAP block: injection of 20ml 0.25% bupvicaine given between internal oblique and transversus abdominis muscle on both sides of midline with no intervention in control group.

VAS (visual analogue score) : VAS , a linear scale that identifies the pain by the self-report of patient, and it is considered as gold standard for evaluation of pain in conscious patients 7. VAS >4 trigger for inj tramadol 1mg/kg i/v.

Analgesic consumption:- postoperative consumption of injection tramadol will be measured within 24hrs after surgery .

HYPOTHESIS:

TAP block is a safe and effective option to control postoperative analgesia after c section by reducing postoperative consumption of opioids.

MATERIALS AND METHODS:

Study design: Randomized control trial Sampling technique: Consecutive non-probability sampling Sample size: Using the study by Uma Srivastava at el, the results of which showed efficacy of TAP block in terms of cumulative tramadol usage during first 24 h after surgery in study group vs control group C as (75 ± 22 vs. 168 ± 45 mg in groups B and C ) and with the help of WHO sample size calculator, following calculations were made Level of significance: 5% Confidence interval: 95% Power of test: 80% Sample size=n= 6 patients in each group As sample size is very small, minimum 30 pts in each group will be used Group A: TAP block will be given Group B: no TAP block will be given Setting: Anesthesia department, Combined Military Hospital, Sargodha ,Pakistan. Duration: After approval from ethical committee Source: Admitted patient Patients will be allocated to two groups A or B, using lottery method. All patients will be assessed on day of surgery and written informed consent will be taken after explaining all the risks and benefits to patient.

On day of surgery, patients will be prepared for surgery and spinal anesthesia as per institutional protocols. Every patient will be given 1.5ml of 0.75% bupivacaine intrathecally to provide anesthesia for c section by consultant anesthetist. During surgery no drug other than oxytocin and anti-emetic (if required) will be given. In group A, at the end of surgery, TAP block will be given via ultrasound guided subcostal approach on both sides of midline. After strict monitoring for next 15-20mins,pt will be shifted to PACU. Time of TAP block will be recorded as time 0.

In ward , all patients will be given analgesia as per departmental protocol (injection ketorolac 30mg i/v TDS).In postoperative period intensity of pain and opioid consumption within 24hrs of surgery will be recorded. Performa till the application of TAP block will be filled by treating anesthetist, whereas remaining will be filled by trainee anesthesia.

After collecting all data, data would be entered and analyzed using SPSS Version 16.

Descriptive statistics will be used to calculate quantitative and qualitative variables. Mean and SD will be calculated for quantitative variables i.e. age weight, intensity of pain, dosage of opioids. Frequency and percentage will be calculated for qualitative variables i.e. gender. P value <0.05 will be considered statistically significant. All results would be presented as frequency tables. Effect modifiers like weight and age will be controlled by stratification and post stratification independent sample t test will be used.

Independent t test will be used to compare group A and B in terms of mean usage of tramadol within 24hrs of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 and 45 years
* Elective cesarean
* Fit to undergo surgery under spinal anesthesia

Exclusion Criteria:

Patients who will have

* Any contraindication to spinal anesthesia
* ASA class III and IV
* Known Allergic to local anesthetic
* Eclampsia
* Placenta accreta/percretra

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-04-25 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
postoperative consumption of opioids | 24hours after surgery
  questionnaire will be filled 24hours after the surgery by trainee anesthesia and he/she will document the total consumption of intravenous tramadol after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Department of Pediatrics, Rawalpindi, Punjab Province
  - Madiha Ahmed, Islamabad

IPD SHARING:
Plan to Share IPD: No